CLINICAL TRIAL: NCT04643834
Title: Validation of Cerebral Non-invasive Monitoring and Prediction of Post-operative Delirium and Outcomes: A Prospective Observational Study
Brief Title: Cerebral Monitoring and Post-operative Delirium and Outcomes
Acronym: Techno-5
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Andre Denault, Principal Investigator, Montreal Heart Institute
Other Study IDs: 2020-2667
Record Dates: First submitted 2020-11-10; First posted 2020-11-25 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Delirium; Cerebral Desaturation; EEG With Abnormally Slow Frequencies
Keywords: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain monitoring using near-infrared spectroscopy (NIRS) started in 2002 in the operating room of the Montreal heart Institute (MHI). This was followed by the use of somatic NIRS in 2010, transcranial Doppler in 2015 and processed electroencephalogram (pEEG) using Sedline (Masimo, Irvine CA) in 2017. The introduction of those modalities led to significant change in intraoperative management. The goal of these devices is to improve our ability to detect and predict post-operative complications as well as offering insights on how to prevent them. The current project explores in further detail the impact of the introduction of pEEG in the operating room and in the intensive care unit (ICU) on post-operative delirium.

DETAILED DESCRIPTION:
Overview of the problem: Post-operative delirium in cardiac surgery Brain monitoring using NIRS started in 2002 in the operating rooms of the MHI. Since that period, the investigators described our experience on 1613 reported patients from published case reports (n=30), cohort studies (n=1270), randomized controlled trials (n=313), and review articles.

In the presence of brain desaturation, the investigators have previously described an algorithmic approach based on a series of interventions (such as head positioning, increasing blood pressure and inspired oxygen etc.) which are triggered by the etiology, one at a time or simultaneously, ideally as early as possible i.e. when the cerebral NIRS value start to decrease by more than 10%. The success rate for correction of brain desaturation was more than 95%.

The use of both cerebral NIRS and pEEG led to new insights which were not apparent when these technologies were used in isolation. For instance, brain desaturation resulting from increased pEEG activity will be observed upon awakening. On the other hand, brain desaturation associated with reduced pEEG activity may indicates brain hypoperfusion. A new algorithm to manage cerebral NIRS and pEEG was introduced and published in May 2019.

This algorithm has not been validated and could represent a major advance in the care of cardiac surgical patients. One of the potential roles of this type of monitoring would be its ability to predict emergence delirium, postoperative delirium and other end-organ complications. Eventually, the early identification could lead to prevention of post-operative complications such as delirium.

Brain oximetry and delirium Between 16% and 30% of elderly hospitalised patients with cardiovascular disease will develop delirium. Delirium and cognitive dysfunction are highly frequent among hospitalized patients across all healthcare settings, but especially in surgical and critical care populations where rates are reported to be as high as 70%. Mortality is increased in patients with delirium after cardiac surgery.

Delirium is defined by the DSM-5 as an acute brain dysfunction associated with attention deficit and altered consciousness. Three types of delirium have been described : hypoactive associated with lethargia, hyperactive with agitation and a combination of both that can alternate. There are several predisposing factors such as pre-operative cognitive dysfunction. A recent systematic review has identified the following factors associated with delirium occurrence. Those factors include advanced age, prior psychiatric condition, mild cognitive impairment, and cerebrovascular disease. Post-operative delirium is associated with prolonged duration of hospitalisation, post-operative complications and increased mortality.

There have been several reports linking reduced cerebral NIRS measurements, delirium and post-operative cognitive dysfunction among surgical populations. The mechanism through which reduced brain saturation and delirium co-exist could include cerebral malperfusion and venous congestion from right heart dysfunction. Those factors have been recently explored and their association with delirium and post-operative cognitive dysfunction has been reported in the ICU as well as in the operating room. As right heart dysfunction can be associated with prolonged period of venous hypertension, this can lead to interstitial edema which can further impairs end organ perfusion such as the brain. In the context of cardiopulmonary bypass (CPB), this phenomenon might be aggravated by alteration in endothelial glycocalyx resulting in increased permeability of the capillary endothelium. The resulting interstitial edema is thought to be a mediator of adverse outcomes in critically ill fluid overloaded patients. In addition to altered NIRS values observed with delirium after cardiac surgery, abnormal brain electrical activity has been described.

Brain electroencephalographic monitoring and delirium Electrical activity of the brain can be monitored through electroencephalography (EEG) and recently bedside monitor of pEEG such as the BIS (Medtronic, USA) or Sedline (Masimo Irvine CA) allow bedside measurement of frontal electrical activity. Delirium is associated with EEG changes, typically global slowing of EEG activity. Significant differences in EEG have been observed in elderly with or without delirium. The alpha, theta and delta wave power and the theta ratio in relation to the other EEG waves are different in patients with or without delirium. Furthermore, significant reduction in EEG activity leading to "burst-suppression" has been related to delirium appearance, prolonged hospital length of stay and mortality. Controversial results have been reported from studies and meta-analysis looking at intervention to correct those factors and improve outcome. However, these observations have never combined information obtained from frontal EEG with brain oximetry. A recent prospective study from Belgium reported an association with post-operative delirium and the information obtained from the combined use of brain NIRS and pEEG.

Previous work of delirium and brain oximetry and electroencephalographic monitoring In 2011, the investigators reported our first experience in the use of NIRS in 61 patients undergoing off-pump bypass cardiac surgery as a predictor post-operative cognitive dysfunction. In 2016, an observational study was conducted with 30 consecutive adults with delirium after cardiac surgery. The mean oximetry value decreased from (mean ± SD) 66.4 ± 6.7 to 50.8 ± 6.8 on the first day after delirium onset and increased in patients whose delirium resorbed over the 3 days. The relationship between oximetry, delirium diagnosis, and severity was analyzed with a marginal model and linear mixed models. Cerebral oximetry was related to delirium diagnosis (p≤.0001) and severity (p≤.0001). In that study, somatic oximetry values were normal in patients with delirium.

The second study, in 2017, was a case-control retrospective study which included 346 patients, of which 39 (11%), 104 (30%), and 142 (41%) patients presented delirium at 24, 48, and 72 hours post-ICU arrival, respectively. The cumulative fluid balance was associated with delirium occurrence (OR 1.20, 95% CI: 1.066-1.355, p=.003). History of neurological disorder, having both hearing and visual impairment, type of procedure, perioperative cerebral oximetry, mean pulmonary artery pressure pre-CPB, and mean arterial pressure post-CPB also contributed to delirium in the model.

In the third study, both a retrospective and prospective cohort were reported including a total of 382 patients. Adult patients who underwent portal venous pulsed-wave Doppler by the attending physician during usual care in the ICU were included in the retrospective cohort (n=237). For the prospective cohort (n=145), patients had a cognitive and echocardiographic evaluation the day before surgery and daily for three days after surgery. Delirium was independently assessed by the nursing staff in the prospective cohort. An association was found between delirium and portal vein pulsatility, a marker of right heart failure, in the retrospective cohort (OR:2.69 CI:1.47-4.90 p=0.001). In the prospective cohort, significant associations were confirmed between the presence of portal vein pulsatility and the development of cognitive dysfunction and asterixis assessed by the investigators (OR:2.10 CI:1.25-3.53 p=0.005 and OR:5.19 [CI:2.27; 11.88] p<0.001) But also the association with delirium detected by the nursing staff was confirmed (HR:2.63 CI:1.13-6.11 p=0.025). Higher NT-pro-BNP measurements (OR:4.03 [CI: 1.78-9.15] p=0.001) and cerebral desaturations (OR:2.54 [CI:1.12-5.76] p=0.03) were associated with cognitive dysfunction. In this third study, baseline daily pEEG were obtained daily in combination with NIRS values. However, no association was observed between delirium and preliminary waveform analysis.

In summary, those studies support an association between episodes of cerebral desaturations measured by brain oximetry and the occurrence of delirium. Venous cerebral congestion as a consequence of right ventricular dysfunction leading to portal hypertension and possibly cytokine release through a cardio-intestinal syndrome appears to be a potential mechanism. As supported by other authors, reduced cerebral NIRS values could be secondary to elevated venous pressure, fluid overload and the latter contribute to a type of congestive delirium. It could also be reflective of increased cerebral metabolism, such as can be observed when patient emerge from general anesthesia after cardiac surgery. However, in those studies, only a single cerebral NIRS and pEEG value were obtained. The combination of both modalities with the use of bilateral cerebral NIRS was not studied prospectively in both the operating room and in the ICU. Currently, it is not known whether the information obtained by these monitors is different in patients presenting an episode of delirium compared to those who do not show any episode of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 18 and older, undergoing cardiac surgery with CPB or off pump CABG

Exclusion Criteria:

* Patient with a critical pre-operative state defined as any of the following: vasopressor requirement, mechanical circulatory support, dialysis, mechanical ventilation, cardiac arrest necessitating resuscitation, aborted sudden death, preoperative cardiac massage, preoperative intra-aortic balloon pump.
* Patient with the diagnosis of delirium at any point before surgery during the current hospitalization
* Emergent surgery
* Surgery under deep hypothermic circulatory arrest

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of neurological events | 72 hours
  Events will be categorized according to change in oxygen saturation measured by near infra-red spectroscopy and according to changes in pEEG activity evaluated by the patient state index, burst suppression ratio and spectral edge frequency. Events will be categorized based on the following classification:
  1. Cerebral desaturation (>10% from baseline) AND a decrease in pEEG activity (patient state index (PSI) < 40 and/or burst suppression ratio (BSR) >0 and/or spectral edge frequency (SEF) <10)
  2. Cerebral desaturation (>10% from baseline) AND an increase in pEEG activity (PSI ≥ 60, BSR = 0, SEF > 15)
  3. Cerebral desaturation (>10% from baseline) AND a normal pEEG activity (PSI ≥ 40-60, BSR = 0 and SEF 10-15)
  4. Normal cerebral saturation (Cerebral desaturation ≤10% from baseline) AND a decrease in pEEG activity (PSI < 40, and/or BSR >0 and/or SEF<10).

SECONDARY OUTCOMES:
Rate of cognitive dysfunction | 72 hours
  Cognitive dysfunction will be defined as a Delirium Index Score ≥1
Rate of delirium | 72 hours
  Delirium will be defined as an Intensive Care Delirium Screening Checklist (ICDSC) : score of ≥4
Duration of persistent organ dysfunction | Up to 28 days or until hospital discharge
  Persistent organ dysfunction is defined as one or more of the following: mechanical ventilation; vasopressor therapy (ongoing need for vasopressor agents such as norepinephrine, epinephrine, vasopressin, dopamine >5 μg/kg/min, or phenylephrine >50 μg/min); mechanical circulatory support (ongoing need for mechanical devices such as ECMO or IABP); new continuous renal replacement therapy or new intermittent hemodialysis (first to last dialysis session). Therefore, TPOD represent the time for which the patient requires invasive life support after cardiac surgery.
  2. ICU stay (in hours) 3. Duration of hospital stay (in days)
Rate of all cause death during hospitalization | Up to 30 days or until hospital discharge
  Death from any cause
Rate of acute kidney injury | Up to 30 days or until hospital discharge
  Defined according to KDIGO serum creatinine criteria: Increase of ≥27 umol/L within 48 hours or ≥50%
Rate of major bleeding | Up to 30 days or until hospital discharge
  Defined by the Bleeding Academic Research Consortium as one of the following:
  Perioperative intracranial bleeding within 48h ii. Reoperation after closure of sternotomy for the purpose of controlling bleeding iii. Transfusion of ≥5 units of whole blood of packed red blood cells within a 48 hours period iv. Chest tube output ≥2L within a 24 hours period.
Rate of surgical re-intervention | Up to 30 days or until hospital discharge
  Second surgery within the same hospitalization for any reason
Rate of stroke | Up to 30 days or until hospital discharge
  Central neurologic deficit persisting longer than 72 hours
Duration of mechanical ventilation | Up to 30 days or until hospital discharge
  Duration of mechanical support with a respirator in an intubated patient

CONTACTS AND LOCATIONS:
Overall Officials: Andre Y Denault, MD, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taillefer MC, Denault AY. Cerebral near-infrared spectroscopy in adult heart surgery: systematic review of its clinical efficacy. Can J Anaesth. 2005 Jan;52(1):79-87. doi: 10.1007/BF03018586. PMID 15625262
- [Background] Denault A, Deschamps A, Murkin JM. A proposed algorithm for the intraoperative use of cerebral near-infrared spectroscopy. Semin Cardiothorac Vasc Anesth. 2007 Dec;11(4):274-81. doi: 10.1177/1089253207311685. PMID 18270192
- [Background] Harel F, Denault A, Ngo Q, Dupuis J, Khairy P. Near-infrared spectroscopy to monitor peripheral blood flow perfusion. J Clin Monit Comput. 2008 Feb;22(1):37-43. doi: 10.1007/s10877-007-9105-9. Epub 2007 Nov 27. PMID 18040873
- [Background] Denault AY, Deschamps A, Couture P. Intraoperative hemodynamic instability during and after separation from cardiopulmonary bypass. Semin Cardiothorac Vasc Anesth. 2010 Sep;14(3):165-82. doi: 10.1177/1089253210376673. Epub 2010 Jul 23. PMID 20656747
- [Background] Denault AY, Haddad F, Jacobsohn E, Deschamps A. Perioperative right ventricular dysfunction. Curr Opin Anaesthesiol. 2013 Feb;26(1):71-81. doi: 10.1097/ACO.0b013e32835b8be2. PMID 23235519
- [Background] Denault AY, Couture P. Practical diastology. World J Anesthesiology. 2014;3(1):96-104
- [Background] St-Pierre P, Deschamps A, Cartier R, Basmadjian AJ, Denault AY. Inhaled milrinone and epoprostenol in a patient with severe pulmonary hypertension, right ventricular failure, and reduced baseline brain saturation value from a left atrial myxoma. J Cardiothorac Vasc Anesth. 2014 Jun;28(3):723-9. doi: 10.1053/j.jvca.2012.10.017. Epub 2013 Apr 26. No abstract available. PMID 23623891
- [Background] Denault A, Lamarche Y, Rochon A, Cogan J, Liszkowski M, Lebon JS, Ayoub C, Taillefer J, Blain R, Viens C, Couture P, Deschamps A. Innovative approaches in the perioperative care of the cardiac surgical patient in the operating room and intensive care unit. Can J Cardiol. 2014 Dec;30(12 Suppl):S459-77. doi: 10.1016/j.cjca.2014.09.029. Epub 2014 Oct 5. PMID 25432139
- [Background] Laflamme M, Perrault LP, Carrier M, Elmi-Sarabi M, Fortier A, Denault AY. Preliminary experience with combined inhaled milrinone and prostacyclin in cardiac surgical patients with pulmonary hypertension. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):38-45. doi: 10.1053/j.jvca.2014.06.012. Epub 2014 Oct 17. PMID 25440627
- [Background] Gebhard CE, Desjardins G, Gebhard C, Gavra P, Denault AY. Intratracheal Milrinone Bolus Administration During Acute Right Ventricular Dysfunction After Cardiopulmonary Bypass. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):489-496. doi: 10.1053/j.jvca.2016.11.033. Epub 2016 Nov 22. PMID 28216201
- [Background] Hu T, Collin Y, Lapointe R, Carrier FM, Massicotte L, Fortier A, Lambert J, Vandenbroucke-Menu F, Denault AY. Preliminary Experience in Combined Somatic and Cerebral Oximetry Monitoring in Liver Transplantation. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):73-84. doi: 10.1053/j.jvca.2017.07.019. Epub 2017 Jul 20. PMID 29229261
- [Background] Lecluyse V, Couture EJ, Denault AY. A Proposed Approach to Cerebral and Somatic Desaturation in the Intensive Care Unit: Preliminary Experience and Review. J Cardiothorac Vasc Anesth. 2017 Oct;31(5):1805-1809. doi: 10.1053/j.jvca.2017.02.175. Epub 2017 Feb 20. No abstract available. PMID 28552296
- [Background] Couture EJ, Provencher S, Denault AY. Management of Severe Pulmonary Hypertensive Disease for Surgical and Nonsurgical Procedures. Int Anesthesiol Clin. 2018 Fall;56(4):e28-e55. doi: 10.1097/AIA.0000000000000202. No abstract available. PMID 30204604
- [Background] Denault AY, Brassard P, Jacquet-Lagreze M, Halwagi AE. Targeting optimal blood pressure monitoring: what's next? J Thorac Dis. 2018 Sep;10(Suppl 26):S3281-S3285. doi: 10.21037/jtd.2018.08.115. No abstract available. PMID 30370138
- [Background] Numan T, van den Boogaard M, Kamper AM, Rood PJT, Peelen LM, Slooter AJC; Dutch Delirium Detection Study Group. Delirium detection using relative delta power based on 1-minute single-channel EEG: a multicentre study. Br J Anaesth. 2019 Jan;122(1):60-68. doi: 10.1016/j.bja.2018.08.021. Epub 2018 Oct 2. PMID 30579407
- [Background] Paquet C, Deschamps A, Denault AY, Couture P, Carrier M, Babin D, Levesque S, Piquette D, Lambert J, Tardif JC. Baseline regional cerebral oxygen saturation correlates with left ventricular systolic and diastolic function. J Cardiothorac Vasc Anesth. 2008 Dec;22(6):840-6. doi: 10.1053/j.jvca.2008.02.013. Epub 2008 May 12. PMID 18834789
- [Background] Gelinas C, Choiniere M, Ranger M, Denault A, Deschamps A, Johnston C. Toward a new approach for the detection of pain in adult patients undergoing cardiac surgery: near-infrared spectroscopy--a pilot study. Heart Lung. 2010 Nov-Dec;39(6):485-93. doi: 10.1016/j.hrtlng.2009.10.018. Epub 2010 Apr 24. PMID 20561850
- [Background] de Tournay-Jette E, Dupuis G, Bherer L, Deschamps A, Cartier R, Denault A. The relationship between cerebral oxygen saturation changes and postoperative cognitive dysfunction in elderly patients after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):95-104. doi: 10.1053/j.jvca.2010.03.019. Epub 2010 Jul 22. PMID 20650659
- [Background] Deschamps A, Denault A, Rochon A, Cogan J, Page P, D'Antono B. Evaluation of autonomic reserves in cardiac surgery patients. J Cardiothorac Vasc Anesth. 2013 Jun;27(3):485-93. doi: 10.1053/j.jvca.2012.07.016. Epub 2012 Oct 1. PMID 23036623
- [Background] Deschamps A, Lambert J, Couture P, Rochon A, Lebon JS, Ayoub C, Cogan J, Denault A. Reversal of decreases in cerebral saturation in high-risk cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1260-6. doi: 10.1053/j.jvca.2013.01.019. Epub 2013 Jun 18. PMID 23791498
- [Background] Mailhot T, Cossette S, Lambert J, Cournoyer A, Denault AY. Cerebral oximetry as a biomarker of postoperative delirium in cardiac surgery patients. J Crit Care. 2016 Aug;34:17-23. doi: 10.1016/j.jcrc.2016.02.024. Epub 2016 Mar 30. PMID 27288603
- [Background] Cournoyer A, Denault A, Cossette S, Fortier A, Daoust R, Iseppon M, Chauny JM, Notebaert E. Reproducibility, interchangeability of measures, time to measure stabilization, and reference values of two tissue oximeters in healthy volunteers. J Biomed Opt. 2016 Sep 1;21(9):97003. doi: 10.1117/1.JBO.21.9.097003. PMID 27637007
- [Background] Eljaiek R, Cavayas YA, Rodrigue E, Desjardins G, Lamarche Y, Toupin F, Denault AY, Beaubien-Souligny W. High postoperative portal venous flow pulsatility indicates right ventricular dysfunction and predicts complications in cardiac surgery patients. Br J Anaesth. 2019 Feb;122(2):206-214. doi: 10.1016/j.bja.2018.09.028. Epub 2018 Nov 28. PMID 30686306
- [Background] Beaubien-Souligny W, Benkreira A, Robillard P, Bouabdallaoui N, Chasse M, Desjardins G, Lamarche Y, White M, Bouchard J, Denault A. Alterations in Portal Vein Flow and Intrarenal Venous Flow Are Associated With Acute Kidney Injury After Cardiac Surgery: A Prospective Observational Cohort Study. J Am Heart Assoc. 2018 Oct 2;7(19):e009961. doi: 10.1161/JAHA.118.009961. PMID 30371304
- [Background] Mailhot T, Cossette S, Lambert J, Beaubien-Souligny W, Cournoyer A, O'Meara E, Maheu-Cadotte MA, Fontaine G, Bouchard J, Lamarche Y, Benkreira A, Rochon A, Denault A. Delirium After Cardiac Surgery and Cumulative Fluid Balance: A Case-Control Cohort Study. J Cardiothorac Vasc Anesth. 2019 Jan;33(1):93-101. doi: 10.1053/j.jvca.2018.07.012. Epub 2018 Aug 17. PMID 30122614
- [Background] Piquette D, Deschamps A, Belisle S, Pellerin M, Levesque S, Tardif JC, Denault AY. Effect of intravenous nitroglycerin on cerebral saturation in high-risk cardiac surgery. Can J Anaesth. 2007 Sep;54(9):718-27. doi: 10.1007/BF03026868. PMID 17766739
- [Background] Denault AY, Bussieres JS, Arellano R, Finegan B, Gavra P, Haddad F, Nguyen AQN, Varin F, Fortier A, Levesque S, Shi Y, Elmi-Sarabi M, Tardif JC, Perrault LP, Lambert J. A multicentre randomized-controlled trial of inhaled milrinone in high-risk cardiac surgical patients. Can J Anaesth. 2016 Oct;63(10):1140-1153. doi: 10.1007/s12630-016-0709-8. Epub 2016 Jul 28. PMID 27470232
- [Background] Deschamps A, Hall R, Grocott H, Mazer CD, Choi PT, Turgeon AF, de Medicis E, Bussieres JS, Hudson C, Syed S, Seal D, Herd S, Lambert J, Denault A, Deschamps A, Mutch A, Turgeon A, Denault A, Todd A, Jerath A, Fayad A, Finnegan B, Kent B, Kennedy B, Cuthbertson BH, Kavanagh B, Warriner B, MacAdams C, Lehmann C, Fudorow C, Hudson C, McCartney C, McIsaac D, Dubois D, Campbell D, Mazer D, Neilpovitz D, Rosen D, Cheng D, Drapeau D, Dillane D, Tran D, Mckeen D, Wijeysundera D, Jacobsohn E, Couture E, de Medicis E, Alam F, Abdallah F, Ralley FE, Chung F, Lellouche F, Dobson G, Germain G, Djaiani G, Gilron I, Hare G, Bryson G, Clarke H, McDonald H, Roman-Smith H, Grocott H, Yang H, Douketis J, Paul J, Beaubien J, Bussieres J, Pridham J, Armstrong JN, Parlow J, Murkin J, Gamble J, Duttchen K, Karkouti K, Turner K, Baghirzada L, Szabo L, Lalu M, Wasowicz M, Bautista M, Jacka M, Murphy M, Schmidt M, Verret M, Perrault MA, Beaudet N, Buckley N, Choi P, MacDougall P, Jones P, Drolet P, Beaulieu P, Taneja R, Martin R, Hall R, George R, Chun R, McMullen S, Beattie S, Sampson S, Choi S, Kowalski S, McCluskey S, Syed S, Boet S, Ramsay T, Saha T, Mutter T, Chowdhury T, Uppal V, Mckay W; Canadian Perioperative Anesthesia Clinical Trials Group. Cerebral Oximetry Monitoring to Maintain Normal Cerebral Oxygen Saturation during High-risk Cardiac Surgery: A Randomized Controlled Feasibility Trial. Anesthesiology. 2016 Apr;124(4):826-36. doi: 10.1097/ALN.0000000000001029. PMID 26808629
- [Background] Hu T, Lavoie A, Deschamps A, Guerra P, Babin D, Fortier A, Lambert J, Denault AY. Can we prevent significant brain desaturation during defibrillator testing by increasing the brain saturation reserve? Can J Anaesth. 2018 Jun;65(6):732-734. doi: 10.1007/s12630-018-1059-5. Epub 2018 Jan 19. No abstract available. PMID 29352417
- [Background] Denault A, Shaaban Ali M, Couture EJ, Beaubien-Souligny W, Bouabdallaoui N, Brassard P, Mailhot T, Jacquet-Lagreze M, Lamarche Y, Deschamps A. A Practical Approach to Cerebro-Somatic Near-Infrared Spectroscopy and Whole-Body Ultrasound. J Cardiothorac Vasc Anesth. 2019 Aug;33 Suppl 1:S11-S37. doi: 10.1053/j.jvca.2019.03.039. PMID 31279350
- [Background] Couture EJ, Deschamps A, Denault AY. Patient management algorithm combining processed electroencephalographic monitoring with cerebral and somatic near-infrared spectroscopy: a case series. Can J Anaesth. 2019 May;66(5):532-539. doi: 10.1007/s12630-019-01305-y. Epub 2019 Feb 1. PMID 30710260
- [Background] Ryan DJ, O'Regan NA, Caoimh RO, Clare J, O'Connor M, Leonard M, McFarland J, Tighe S, O'Sullivan K, Trzepacz PT, Meagher D, Timmons S. Delirium in an adult acute hospital population: predictors, prevalence and detection. BMJ Open. 2013 Jan 7;3(1):e001772. doi: 10.1136/bmjopen-2012-001772. PMID 23299110
- [Background] McPherson JA, Wagner CE, Boehm LM, Hall JD, Johnson DC, Miller LR, Burns KM, Thompson JL, Shintani AK, Ely EW, Pandharipande PP. Delirium in the cardiovascular ICU: exploring modifiable risk factors. Crit Care Med. 2013 Feb;41(2):405-13. doi: 10.1097/CCM.0b013e31826ab49b. PMID 23263581
- [Background] Giuseffi JL, Borges N, Boehm L, Wang L, McPherson J, Fredi J, et al. DELIRIUM AND TRANSCATHETER AORTIC VALVE REPLACEMENT. J Am Coll Cardiol. 2014;63(12):A1736
- [Background] Honda S, Nagai T, Sugano Y, Okada A, Asaumi Y, Aiba T, Noguchi T, Kusano K, Ogawa H, Yasuda S, Anzai T; NaDEF investigators. Prevalence, determinants, and prognostic significance of delirium in patients with acute heart failure. Int J Cardiol. 2016 Nov 1;222:521-527. doi: 10.1016/j.ijcard.2016.07.236. Epub 2016 Jul 30. PMID 27509220
- [Background] Grotti S, Falsini G. Delirium in cardiac patients. Eur Heart J. 2017 Aug 1;38(29):2244. doi: 10.1093/eurheartj/ehx380. No abstract available. PMID 28810719
- [Background] Mailhot T, Cossette S, Cote J, Bourbonnais A, Cote MC, Lamarche Y, Denault A. A post cardiac surgery intervention to manage delirium involving families: a randomized pilot study. Nurs Crit Care. 2017 Jul;22(4):221-228. doi: 10.1111/nicc.12288. Epub 2017 Mar 31. PMID 28371230
- [Background] Sockalingam S, Parekh N, Bogoch II, Sun J, Mahtani R, Beach C, Bollegalla N, Turzanski S, Seto E, Kim J, Dulay P, Scarrow S, Bhalerao S. Delirium in the postoperative cardiac patient: a review. J Card Surg. 2005 Nov-Dec;20(6):560-7. doi: 10.1111/j.1540-8191.2005.00134.x. PMID 16309412
- [Background] Gottesman RF, Grega MA, Bailey MM, Pham LD, Zeger SL, Baumgartner WA, Selnes OA, McKhann GM. Delirium after coronary artery bypass graft surgery and late mortality. Ann Neurol. 2010 Mar;67(3):338-44. doi: 10.1002/ana.21899. PMID 20373345
- [Background] Association AP. Diagnostic and Statistical Manual of Mental Disorders: Dsm-5: Amer Psychiatric Pub Incorporated; 2013
- [Background] Rudolph JL, Marcantonio ER. Review articles: postoperative delirium: acute change with long-term implications. Anesth Analg. 2011 May;112(5):1202-11. doi: 10.1213/ANE.0b013e3182147f6d. Epub 2011 Apr 7. PMID 21474660
- [Background] Fick DM, Mion LC. How to try this: Delirium superimposed on dementia. Am J Nurs. 2008 Jan;108(1):52-60; quiz 61. doi: 10.1097/01.NAJ.0000304476.80530.7d. PMID 18156861
- [Background] Fick DM, Steis MR, Waller JL, Inouye SK. Delirium superimposed on dementia is associated with prolonged length of stay and poor outcomes in hospitalized older adults. J Hosp Med. 2013 Sep;8(9):500-5. doi: 10.1002/jhm.2077. Epub 2013 Aug 19. PMID 23955965
- [Background] Gosselt AN, Slooter AJ, Boere PR, Zaal IJ. Risk factors for delirium after on-pump cardiac surgery: a systematic review. Crit Care. 2015 Sep 23;19(1):346. doi: 10.1186/s13054-015-1060-0. PMID 26395253
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Madsen PL, Nielsen HB, Christiansen P. Well-being and cerebral oxygen saturation during acute heart failure in humans. Clin Physiol. 2000 Mar;20(2):158-64. doi: 10.1046/j.1365-2281.2000.00241.x. PMID 10735984
- [Background] Madsen PL, Secher NH. Postoperative confusion preceded by decreased frontal lobe haemoglobin oxygen saturation. Anaesth Intensive Care. 2000 Jun;28(3):308-10. doi: 10.1177/0310057X0002800310. PMID 10853215
- [Background] Edmonds HL, Jr., Cao L, Yu QJ. In the elderly, coronary artery bypass grafting associated with more brain O2 desaturation and cognitive dysfunction. The Annals of thoracic surgery. 2002;73:S375
- [Background] Hong SW, Shim JK, Choi YS, Kim DH, Chang BC, Kwak YL. Prediction of cognitive dysfunction and patients' outcome following valvular heart surgery and the role of cerebral oximetry. Eur J Cardiothorac Surg. 2008 Apr;33(4):560-5. doi: 10.1016/j.ejcts.2008.01.012. Epub 2008 Feb 12. PMID 18272385
- [Background] Pfister D, Siegemund M, Dell-Kuster S, Smielewski P, Ruegg S, Strebel SP, Marsch SC, Pargger H, Steiner LA. Cerebral perfusion in sepsis-associated delirium. Crit Care. 2008;12(3):R63. doi: 10.1186/cc6891. Epub 2008 May 5. PMID 18457586
- [Background] Morimoto Y, Yoshimura M, Utada K, Setoyama K, Matsumoto M, Sakabe T. Prediction of postoperative delirium after abdominal surgery in the elderly. J Anesth. 2009;23(1):51-6. doi: 10.1007/s00540-008-0688-1. Epub 2009 Feb 22. PMID 19234823
- [Background] Brady K, Joshi B, Zweifel C, Smielewski P, Czosnyka M, Easley RB, Hogue CW Jr. Real-time continuous monitoring of cerebral blood flow autoregulation using near-infrared spectroscopy in patients undergoing cardiopulmonary bypass. Stroke. 2010 Sep;41(9):1951-6. doi: 10.1161/STROKEAHA.109.575159. Epub 2010 Jul 22. PMID 20651274
- [Background] Brady KM, Mytar JO, Lee JK, Cameron DE, Vricella LA, Thompson WR, Hogue CW, Easley RB. Monitoring cerebral blood flow pressure autoregulation in pediatric patients during cardiac surgery. Stroke. 2010 Sep;41(9):1957-62. doi: 10.1161/STROKEAHA.109.575167. Epub 2010 Jul 22. PMID 20651273
- [Background] Schoen J, Meyerrose J, Paarmann H, Heringlake M, Hueppe M, Berger KU. Preoperative regional cerebral oxygen saturation is a predictor of postoperative delirium in on-pump cardiac surgery patients: a prospective observational trial. Crit Care. 2011;15(5):R218. doi: 10.1186/cc10454. Epub 2011 Sep 19. PMID 21929765
- [Background] Siepe M, Pfeiffer T, Gieringer A, Zemann S, Benk C, Schlensak C, Beyersdorf F. Increased systemic perfusion pressure during cardiopulmonary bypass is associated with less early postoperative cognitive dysfunction and delirium. Eur J Cardiothorac Surg. 2011 Jul;40(1):200-7. doi: 10.1016/j.ejcts.2010.11.024. Epub 2010 Dec 18. PMID 21168339
- [Background] Palmbergen WA, van Sonderen A, Keyhan-Falsafi AM, Keunen RW, Wolterbeek R. Improved perioperative neurological monitoring of coronary artery bypass graft patients reduces the incidence of postoperative delirium: the Haga Brain Care Strategy. Interact Cardiovasc Thorac Surg. 2012 Oct;15(4):671-7. doi: 10.1093/icvts/ivs317. Epub 2012 Jul 9. PMID 22778141
- [Background] Papadopoulos G, Karanikolas M, Liarmakopoulou A, Papathanakos G, Korre M, Beris A. Cerebral oximetry and cognitive dysfunction in elderly patients undergoing surgery for hip fractures: a prospective observational study. Open Orthop J. 2012;6:400-5. doi: 10.2174/1874325001206010400. Epub 2012 Sep 3. PMID 22962570
- [Background] Lin R, Zhang F, Xue Q, Yu B. Accuracy of regional cerebral oxygen saturation in predicting postoperative cognitive dysfunction after total hip arthroplasty: regional cerebral oxygen saturation predicts POCD. J Arthroplasty. 2013 Mar;28(3):494-7. doi: 10.1016/j.arth.2012.06.041. Epub 2012 Nov 12. PMID 23151365
- [Background] Zheng F, Sheinberg R, Yee MS, Ono M, Zheng Y, Hogue CW. Cerebral near-infrared spectroscopy monitoring and neurologic outcomes in adult cardiac surgery patients: a systematic review. Anesth Analg. 2013 Mar;116(3):663-76. doi: 10.1213/ANE.0b013e318277a255. Epub 2012 Dec 24. PMID 23267000
- [Background] Hori D, Brown C, Ono M, Rappold T, Sieber F, Gottschalk A, Neufeld KJ, Gottesman R, Adachi H, Hogue CW. Arterial pressure above the upper cerebral autoregulation limit during cardiopulmonary bypass is associated with postoperative delirium. Br J Anaesth. 2014 Dec;113(6):1009-17. doi: 10.1093/bja/aeu319. Epub 2014 Sep 25. PMID 25256545
- [Background] Choi JW, Joo Ahn H, Yang M, Kim JA, Lee SM, Ahn JH. Comparison Between Phenylephrine and Dopamine in Maintaining Cerebral Oxygen Saturation in Thoracic Surgery: A Randomized Controlled Trial. Medicine (Baltimore). 2015 Dec;94(49):e2212. doi: 10.1097/MD.0000000000002212. PMID 26656357
- [Background] Colak Z, Borojevic M, Bogovic A, Ivancan V, Biocina B, Majeric-Kogler V. Influence of intraoperative cerebral oximetry monitoring on neurocognitive function after coronary artery bypass surgery: a randomized, prospective study. Eur J Cardiothorac Surg. 2015 Mar;47(3):447-54. doi: 10.1093/ejcts/ezu193. Epub 2014 May 7. PMID 24810757
- [Background] Kara I, Erkin A, Sacli H, Demirtas M, Percin B, Diler MS, Kirali K. The Effects of Near-Infrared Spectroscopy on the Neurocognitive Functions in the Patients Undergoing Coronary Artery Bypass Grafting with Asymptomatic Carotid Artery Disease: A Randomized Prospective Study. Ann Thorac Cardiovasc Surg. 2015;21(6):544-50. doi: 10.5761/atcs.oa.15-00118. Epub 2015 Jun 30. PMID 26133933
- [Background] Trafidlo T, Gaszynski T, Gaszynski W, Nowakowska-Domagala K. Intraoperative monitoring of cerebral NIRS oximetry leads to better postoperative cognitive performance: a pilot study. Int J Surg. 2015 Apr;16(Pt A):23-30. doi: 10.1016/j.ijsu.2015.02.009. Epub 2015 Feb 18. PMID 25701620
- [Background] Hori D, Max L, Laflam A, Brown C, Neufeld KJ, Adachi H, Sciortino C, Conte JV, Cameron DE, Hogue CW Jr, Mandal K. Blood Pressure Deviations From Optimal Mean Arterial Pressure During Cardiac Surgery Measured With a Novel Monitor of Cerebral Blood Flow and Risk for Perioperative Delirium: A Pilot Study. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):606-12. doi: 10.1053/j.jvca.2016.01.012. Epub 2016 Jan 12. PMID 27321787
- [Background] Cerebral Oxygenation and Neurological Outcomes Following Critical Illness (CONFOCAL) Research Group; Canadian Critical Care Trials Group; Wood MD, Maslove DM, Muscedere JG, Day AG, Gordon Boyd J. Low brain tissue oxygenation contributes to the development of delirium in critically ill patients: A prospective observational study. J Crit Care. 2017 Oct;41:289-295. doi: 10.1016/j.jcrc.2017.06.009. Epub 2017 Jun 15. PMID 28668768
- [Background] Haggstrom L, Welschinger R, Caplan GA. Functional neuroimaging offers insights into delirium pathophysiology: A systematic review. Australas J Ageing. 2017 Sep;36(3):186-192. doi: 10.1111/ajag.12417. Epub 2017 May 18. PMID 28519903
- [Background] Lei L, Katznelson R, Fedorko L, Carroll J, Poonawala H, Machina M, Styra R, Rao V, Djaiani G. Cerebral oximetry and postoperative delirium after cardiac surgery: a randomised, controlled trial. Anaesthesia. 2017 Dec;72(12):1456-1466. doi: 10.1111/anae.14056. Epub 2017 Sep 22. PMID 28940368
- [Background] Lopez MG, Pandharipande P, Morse J, Shotwell MS, Milne GL, Pretorius M, Shaw AD, Roberts LJ 2nd, Billings FT 4th. Intraoperative cerebral oxygenation, oxidative injury, and delirium following cardiac surgery. Free Radic Biol Med. 2017 Feb;103:192-198. doi: 10.1016/j.freeradbiomed.2016.12.039. Epub 2016 Dec 27. PMID 28039082
- [Background] Rogers CA, Stoica S, Ellis L, Stokes EA, Wordsworth S, Dabner L, Clayton G, Downes R, Nicholson E, Bennett S, Angelini GD, Reeves BC, Murphy GJ. Randomized trial of near-infrared spectroscopy for personalized optimization of cerebral tissue oxygenation during cardiac surgery. Br J Anaesth. 2017 Sep 1;119(3):384-393. doi: 10.1093/bja/aex182. PMID 28969313
- [Background] Zorrilla-Vaca A, Healy R, Grant MC, Joshi B, Rivera-Lara L, Brown C, Mirski MA. Intraoperative cerebral oximetry-based management for optimizing perioperative outcomes: a meta-analysis of randomized controlled trials. Can J Anaesth. 2018 May;65(5):529-542. doi: 10.1007/s12630-018-1065-7. Epub 2018 Jan 18. PMID 29427259
- [Background] Momeni M, Meyer S, Docquier MA, Lemaire G, Kahn D, Khalifa C, Rosal Martins M, Van Dyck M, Jacquet LM, Peeters A, Watremez C. Predicting postoperative delirium and postoperative cognitive decline with combined intraoperative electroencephalogram monitoring and cerebral near-infrared spectroscopy in patients undergoing cardiac interventions. J Clin Monit Comput. 2019 Dec;33(6):999-1009. doi: 10.1007/s10877-019-00253-8. Epub 2019 Jan 11. PMID 30635867
- [Background] Benkreira A, Beaubien-Souligny W, Mailhot T, Bouabdallaoui N, Robillard P, Desjardins G, Lamarche Y, Cossette S, Denault A. Portal Hypertension Is Associated With Congestive Encephalopathy and Delirium After Cardiac Surgery. Can J Cardiol. 2019 Sep;35(9):1134-1141. doi: 10.1016/j.cjca.2019.04.006. Epub 2019 Apr 16. PMID 31395469
- [Background] Ameloot K, Genbrugge C, Meex I, Eertmans W, Jans F, De Deyne C, Dens J, Mullens W, Ferdinande B, Dupont M. Is venous congestion associated with reduced cerebral oxygenation and worse neurological outcome after cardiac arrest? Crit Care. 2016 May 15;20(1):146. doi: 10.1186/s13054-016-1297-2. PMID 27179510
- [Background] Svennevig K, Hoel T, Thiara A, Kolset S, Castelheim A, Mollnes T, Brosstad F, Fosse E, Svennevig J. Syndecan-1 plasma levels during coronary artery bypass surgery with and without cardiopulmonary bypass. Perfusion. 2008 May;23(3):165-71. doi: 10.1177/0267659108098215. PMID 19029267
- [Background] Bruegger D, Brettner F, Rossberg I, Nussbaum C, Kowalski C, Januszewska K, Becker BF, Chappell D. Acute degradation of the endothelial glycocalyx in infants undergoing cardiac surgical procedures. Ann Thorac Surg. 2015 Mar;99(3):926-31. doi: 10.1016/j.athoracsur.2014.10.013. Epub 2015 Jan 17. PMID 25601655
- [Background] Koning NJ, Vonk AB, Vink H, Boer C. Side-by-Side Alterations in Glycocalyx Thickness and Perfused Microvascular Density During Acute Microcirculatory Alterations in Cardiac Surgery. Microcirculation. 2016 Jan;23(1):69-74. doi: 10.1111/micc.12260. PMID 26638697
- [Background] Glassford NJ, Gelbart B, Bellomo R. Coming full circle: thirty years of paediatric fluid resuscitation. Anaesth Intensive Care. 2017 May;45(3):308-319. doi: 10.1177/0310057X1704500306. PMID 28486889
- [Background] van der Kooi AW, Zaal IJ, Klijn FA, Koek HL, Meijer RC, Leijten FS, Slooter AJ. Delirium detection using EEG: what and how to measure. Chest. 2015 Jan;147(1):94-101. doi: 10.1378/chest.13-3050. PMID 25166725
- [Background] van der Kooi AW, Leijten FS, van der Wekken RJ, Slooter AJ. What are the opportunities for EEG-based monitoring of delirium in the ICU? J Neuropsychiatry Clin Neurosci. 2012 Fall;24(4):472-7. doi: 10.1176/appi.neuropsych.11110347. PMID 23224454
- [Background] Palanca BJA, Wildes TS, Ju YS, Ching S, Avidan MS. Electroencephalography and delirium in the postoperative period. Br J Anaesth. 2017 Aug 1;119(2):294-307. doi: 10.1093/bja/aew475. PMID 28854540
- [Background] Fleischmann R, Trankner S, Bathe-Peters R, Ronnefarth M, Schmidt S, Schreiber SJ, Brandt SA. Diagnostic Performance and Utility of Quantitative EEG Analyses in Delirium: Confirmatory Results From a Large Retrospective Case-Control Study. Clin EEG Neurosci. 2019 Mar;50(2):111-120. doi: 10.1177/1550059418767584. Epub 2018 Apr 10. PMID 29631447
- [Background] Sessler DI, Sigl JC, Kelley SD, Chamoun NG, Manberg PJ, Saager L, Kurz A, Greenwald S. Hospital stay and mortality are increased in patients having a "triple low" of low blood pressure, low bispectral index, and low minimum alveolar concentration of volatile anesthesia. Anesthesiology. 2012 Jun;116(6):1195-203. doi: 10.1097/ALN.0b013e31825683dc. PMID 22546967
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235
- [Background] Kertai MD, White WD, Gan TJ. Cumulative duration of "triple low" state of low blood pressure, low bispectral index, and low minimum alveolar concentration of volatile anesthesia is not associated with increased mortality. Anesthesiology. 2014 Jul;121(1):18-28. doi: 10.1097/ALN.0000000000000281. PMID 24936920
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] MacKenzie KK, Britt-Spells AM, Sands LP, Leung JM. Processed Electroencephalogram Monitoring and Postoperative Delirium: A Systematic Review and Meta-analysis. Anesthesiology. 2018 Sep;129(3):417-427. doi: 10.1097/ALN.0000000000002323. PMID 29912008
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Background] Dabrowski W, Kotlinska E, Rzecki Z, Czajkowski M, Stadnik A, Olszewski K. Raised jugular venous pressure intensifies release of brain injury biomarkers in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):999-1006. doi: 10.1053/j.jvca.2012.07.015. PMID 23122298
- [Background] Kotlinska-Hasiec E, Czajkowski M, Rzecki Z, Stadnik A, Olszewski K, Rybojad B, Dabrowski W. Disturbance in venous outflow from the cerebral circulation intensifies the release of blood-brain barrier injury biomarkers in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):328-35. doi: 10.1053/j.jvca.2013.05.008. Epub 2013 Sep 26. PMID 24075637
- [Background] Lahiri S, Schlick KH, Padrick MM, Rinsky B, Gonzalez N, Jones H, Mayer SA, Lyden PD. Cerebral Pulsatility Index Is Elevated in Patients with Elevated Right Atrial Pressure. J Neuroimaging. 2018 Jan;28(1):95-98. doi: 10.1111/jon.12456. Epub 2017 Jul 3. PMID 28670797
- [Background] Nguyen DN, Huyghens L, Parra J, Schiettecatte J, Smitz J, Vincent JL. Hypotension and a positive fluid balance are associated with delirium in patients with shock. PLoS One. 2018 Aug 7;13(8):e0200495. doi: 10.1371/journal.pone.0200495. eCollection 2018. PMID 30086136
- [Background] Heyland DK, Muscedere J, Drover J, Jiang X, Day AG; Canadian Critical Care Trials Group. Persistent organ dysfunction plus death: a novel, composite outcome measure for critical care trials. Crit Care. 2011;15(2):R98. doi: 10.1186/cc10110. Epub 2011 Mar 18. PMID 21418560
- [Background] Stoppe C, McDonald B, Benstoem C, Elke G, Meybohm P, Whitlock R, Fremes S, Fowler R, Lamarche Y, Jiang X, Day AG, Heyland DK. Evaluation of Persistent Organ Dysfunction Plus Death As a Novel Composite Outcome in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):30-8. doi: 10.1053/j.jvca.2015.07.035. Epub 2015 Jul 29. PMID 26847748
- [Background] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 1--coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S2-22. doi: 10.1016/j.athoracsur.2009.05.053. PMID 19559822
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the Nomenclature of Cognitive Change Associated with Anaesthesia and Surgery-2018. Anesthesiology. 2018 Nov;129(5):872-879. doi: 10.1097/ALN.0000000000002334. PMID 30325806
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Nashef SA, Roques F, Sharples LD, Nilsson J, Smith C, Goldstone AR, Lockowandt U. EuroSCORE II. Eur J Cardiothorac Surg. 2012 Apr;41(4):734-44; discussion 744-5. doi: 10.1093/ejcts/ezs043. Epub 2012 Feb 29. PMID 22378855
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473